CLINICAL TRIAL: NCT00002357
Title: A Multicenter, Randomized, Double-Blinded, Dose-Escalation Study Evaluating the Safety and Antiretroviral Activity of HBY 097 Versus HBY 097 Plus AZT in Patients With Asymptomatic or Mildly Symptomatic HIV Infection
Brief Title: The Safety and Effectiveness of HBY 097 Used With or Without AZT in HIV-Infected Patients Who Have Mild or No Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoechst Marion Roussel (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 252A; HBY097/2001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-05

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; AIDS-Related Complex; Antiviral Agents; Zidovudine
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — HBY 097; Zidovudine

INTERVENTIONS:
Drug: HBY 097
Drug: Zidovudine

SUMMARY:
To obtain preliminary information on the safety, tolerability, and antiretroviral activity of HBY 097 alone or in combination with zidovudine ( AZT ) versus AZT alone.

PER 1/19/96 AMENDMENT: AZT monotherapy arm was eliminated.

DETAILED DESCRIPTION:
Patients are randomized to receive one of three doses of HBY 097 with or without AZT or AZT alone for 12 weeks (AZT monotherapy arm eliminated per 1/19/96 amendment). All patients at a given dose level of HBY 097 must be enrolled and adequate safety data obtained before escalation in subsequent patients begins. Additional patients are entered at the optimal dose of HBY 097. Patients are evaluated weekly for the first 4 weeks and then every 2 weeks for the next 9 weeks.

PER AMENDMENT: Enrollment to the lowest dose cohort is completed.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Treatment for opportunistic infection that develops on study.

Recommended:

* PCP prophylaxis if CD4 count falls below 200 cells/mm3.

Patients must have:

* HIV infection.
* CD4 count 200 - 500 cells/mm3.
* HIV-1 RNA PCR value of 10000 copies/ml or higher.
* Asymptomatic or mildly symptomatic disease.
* No past or current AIDS-defining event.
* Consent of parent or guardian if less than legal age of consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Endocrine, hepatic, renal, or gastrointestinal disease.
* Cardiovascular conduction disease.
* Concomitant medical illness that may complicate study conduct or interpretation of results.
* Other factors that may interfere with patient compliance.

Concurrent Medication:

Excluded:

* Antiretroviral agents other than study drugs.
* Oral contraceptives.
* Cytotoxic chemotherapy.
* Immunomodulators.
* Antiproliferative agents.
* Corticosteroids.
* Anabolic steroids.
* Estrogens.
* Quinoxaline derivatives.

Concurrent Treatment:

Excluded:

* Radiation therapy.

Patients with the following prior conditions are excluded:

* History of hypersensitivity to quinoxaline derivatives or intolerance to AZT.
* History of cardiovascular conduction disease.
* Prior participation in this study or any study using HBY 097.
* Recent use of a drug that interferes with drug metabolism, absorption, distribution, or excretion.
* History of thyroid disease.

Prior Medication:

Excluded at any time:

Prior non-nucleoside reverse transcriptase inhibitors.

Excluded within 30 days prior to study entry:

* Any antiretroviral therapy.
* Oral contraceptives.
* Immunomodulating agents such as systemic corticosteroids, interleukins, or interferons.
* Cytotoxic chemotherapeutic agents.
* Other investigational drugs.

Excluded within 6 months prior to study entry:

Immunotherapeutic vaccine.

Prior Treatment:

Excluded within 30 days prior to study entry:

* Radiation therapy.
* An experimental device. Current ethanol or illicit drug abuse.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Stanford Univ School of Medicine, Stanford, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Med College of Georgia, Augusta, Georgia
  - New York Univ Med Ctr, New York, New York
  - Houston Clinical Research Network, Houston, Texas